CLINICAL TRIAL: NCT04028440
Title: Preliminary Exploration of γδT Cells Immunotherapy in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL).
Brief Title: γδT Cells Immunotherapy in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Beijing GD Initiative Cell Therapy Technology Co., Ltd. (Industry); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zou Dehui, Chief physician, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT2019001-EC-2
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-07

CONDITIONS: Non-Hodgkin's Lymphoma; Relapsed or Refractory B Cell Non-Hodgkin's Lymphoma; Chronic Lymphoblastic Leukemia; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: Biological: Autologous γδT cells Cells will be extracted by apheresis, followed by expanding and activating. The autologous γδT cells product will be adoptive transferred.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous γδT cells (Experimental): Subjects will receive 3 cycles of γδT cells treatments, at four-week intervals, each cycle has 2 infusions, single infusion intravenously at a target dose of 1~2×10e9 γδT cells (constant dose).
  Interventions: Biological: Autologous γδT cells

INTERVENTIONS:
Biological: Autologous γδT cells — Cells will be extracted by apheresis, followed by expanding and activating. The autologous γδT cells product will be adoptive transferred.

SUMMARY:
This study aims to evaluate the safety and efficacy of autologous γδT cells in patients with relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL), chronic lymphoblastic leukemia (CLL) and peripheral T cell lymphoma (PTCL) expect for γδT lymphoma.

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, open label, no control, prospective clinical trial. The study will include the following sequential phases: sign informed consent, γδT cells pre-culture, screening and registration to the trial, apheresis, γδT cells preparation, pre-treatment for lymphodepleting chemotherapy (selectable plan), treatment and follow-up. The study will evaluate the safety and efficacy of the autologous γδT cells in patients with relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL), chronic lymphoblastic leukemia (CLL) and peripheral T cell lymphoma (PTCL) expect for γδT lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should sign informed consent form voluntarily.
2. Gender unlimited, age ≥ 18 years old.
3. Patients with relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL), chronic lymphoblastic leukemia (CLL) and peripheral T cell lymphoma(PTCL) expect for γδT lymphoma.
4. Patients had an evaluable imaging lesion of at least greater than 1.5 cm (except CLL).
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
6. Adequate bone marrow function as defined by：Absolute neutrophil count (ANC) >1000/mm3；Absolute lymphocyte count (ALC) ≥300/mm3；Platelet ≥50000/mm3；Hemoglobin >8.0g/dl.
7. Adequate end organ function as defined by: Total bilirubin ≤ 2 x upper limit of normal（ULN）; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN; Creatinine ≤ 1.5 x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of ≥ 60ml/min.
8. Male and female of reproductive potential must agree to use birth control during the study and for at least 6 weeks post study.

Exclusion Criteria:

1. Patients with history of allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
2. Active central nervous system (CNS) lymphoma; Patients with symptoms of CNS disease must undergo lumbar puncture and brain nuclear magnetic resonance to exclude CNS lymphoma.
3. Patients receiving chemotherapy within 2 weeks prior to γδT cell infusion, with the following exceptions:

   * Pretreatment chemotherapy prescribed by the protocol
   * In order to prevent CNS intrathecal chemotherapy (should be stopped 1 week before γδT cell therapy)
   * Other exploratory combined medications
4. Patients with systemic vasculitis, or with active or uncontrolled autoimmune diseases, as well as primary or secondary immunodeficiency diseases.
5. Active chronic hepatitis B or hepatitis C virus infection, active cytomegalovirus (CMV), EBV infection.
6. Major surgery that was evaluated by the investigator as unsuitable for inclusion within 4 weeks prior to screening.
7. History of other malignant tumors, with the following exceptions

   * Excisional non-melanoma (e.g. cutaneous basal cell carcinoma)
   * Cured situ carcinoma (e.g. cervical carcinoma)
   * Localized prostate cancer with radiotherapy or surgery
   * Patients with a history of malignant tumors, but the disease has been cured for ≥2 years
8. Patient's cardiac function meets any of the following conditions

   * Left ventricular ejection fraction (LVEF) ≤45%
   * Class III or IV heart failure according to the NYHA Heart Failure Classifications
   * QTcB>450 msec
   * Other cardiac disease that investigators judge is not suitable for enrollment
9. History of epilepsy or other active central nervous system disorders.
10. Inoculated live vaccine within 6 weeks before screening.
11. Uncontrolled serious active infection (such as sepsis, bacteremia and fungemia).
12. Patients are allergic to cytokines.
13. Expected survival < 12 weeks.
14. Participated in any other interventional clinical trial within three months.
15. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety. | 15 months
  Incidence of adverse events (AEs) and serious adverse events (SAEs) of each patient will be recorded and analyzed.
Overall response rate (ORR) | 28 days after infusion of γδT cells
  Rate of complete remission (CR) and partial remission (PR).

SECONDARY OUTCOMES:
Duration of remission (DOR) | 15 months
  Duration of remission is defined as the time from the first occurrence of CR or PR in the tumor assessment to the first occurrence of disease progression (PD) or death.
Time to response(TTR) | 15 months
  Time to response is defined as the time from the first administration of trial drug to the first occurrence of CR or PR in the tumor assessment.
Disease control rate (DCR) | 15 months
  Disease control rate is defined as the proportion of subjects who achieved CR, PR, and disease stability (SD) by imaging evaluation.
Progression free survival (PFS) | 15 months
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause.
Overall survival (OS) | 15 months
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Disease Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No